CLINICAL TRIAL: NCT00411970
Title: 20- Versus 23- Gauge System for Pars Plana Vitrectomy: A Prospective Randomized Clinical Study
Brief Title: 20- Versus 23- Gauge System for Pars Plana Vitrectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Ludwig Boltzmann Institute of Retinology and Biomicroscopic Laser Surgery (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23 versus 20 gauge
Record Dates: First submitted 2006-12-14; First posted 2006-12-15 (Estimated); Last update posted 2007-10-25 (Estimated); Status verified 2007-10

CONDITIONS: Diabetic Retinopathy; Macular Edema; Postoperative Complications; Vitreous Hemorrhage
Keywords: 23 gauge pars plana vitrectomy; conjunctival erythema and injection; 20 gauge pars plana vitrectomy; vitreous and retinal surgery
MeSH Terms: conditions — Diabetic Retinopathy; Macular Edema; Postoperative Complications; Vitreous Hemorrhage

INTERVENTIONS:
Device: 20- and 23 gauge vitreoretinal surgery systems

SUMMARY:
The aim of the present study is to compare the functional and clinical differences and advantages between a standard operating system and a newly developed even smaller system for pars plana vitrectomy.

The present study may work out the possible advantages and disadvantages between the routinely used 20-gauge vitrectomy system and the newly developed 23-gauge device.

DETAILED DESCRIPTION:
60 patient randomized into 2 groups of 30 each. All of them operated in general anesthesia, vitrectomized and cataract extracted by phacoemulsification if indicated. Preoperative and postoper5ative controls at days 1,2,3 and week 1, month 1,3 and 12 performed. Parameters of interest are: postoperative conjunctival injection, pain, eye pressure, complications intra- and postoperative as well as the durations of surgery divided into opening time, vitrectomy time, retinal manipulation time, closing time.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Written form of consent
* Vitreous and retinal pathologies requiring surgery

Exclusion Criteria:

* Previous history of vitreous or retinal surgery
* Pregnant or breastfeeding women
* Prohibiting general medical conditions or diseases
* No informed consent signed
* Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2004-09; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Conjunctival Injection
Subjective postoperative recovery

SECONDARY OUTCOMES:
Surgery time
Intraocular pressure
Visual acuity
Technically successful surgery (from surgeon's view)
Intra- and postoperative complications

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Binder, Prof. MD, Principal Investigator — Ludwig Boltzmann Institute for Retinology and Biomicroscopic Laser Surgery; Lukas M Kellner, MD, Study Director — Ludwig Boltzmann Institute for Retinology and Biomicroscopic Laser Surgery; Barbara Wimpissinger, MD, Study Chair — Ludwig Boltzmann Institute for Retinology and Biomicroscopic Laser Surgery
Locations (1):
- Ludwig Boltzmann Institute for Retinology and Biomicroscopic Laser Surgery, Vienna, Austria